CLINICAL TRIAL: NCT05735483
Title: A Phase 3, Multicenter, Long-Term Extension Study to Assess the Safety and Efficacy of Lebrikizumab in Participants 6 Months to <18 Years of Age With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study to Assess the Long-Term Safety and Efficacy of Lebrikizumab (LY3650150) in Participants 6 Months to <18 Years of Age With Moderate-to-Severe Atopic Dermatitis
Acronym: ADorable-2
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18266; J2T-MC-KGBJ/DRM06-AD16 (Other: Eli Lilly and Company); 2022-501478-21-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — lebrikizumab

STUDY DESIGN:
Masking Description: All participants receive Lebrikizumab during the 16-week blinded treatment period. At Week 18, participants receive open-label lebrikizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lebrikizumab (Experimental): Participants will receive Lebrikizumab administered subcutaneously (SC).
  Placebo will be administered to maintain the blind of parent study J2T-MC-KGBI.
  Interventions: Drug: Lebrikizumab; Drug: Placebo
- Lebrikizumab - Optional Extension Period (OEP) (Experimental): During the OEP, participants will be assigned to dose and treatment group based on participant weight and response achieved at treatment week-52.
  Interventions: Drug: Lebrikizumab

INTERVENTIONS:
Drug: Lebrikizumab — Administered SC
  Other Names: LY3650150
Drug: Placebo — Administered SC
  Arms: Lebrikizumab

SUMMARY:
The main purpose of this study is to assess the long-term safety and efficacy of lebrikizumab in participants 6 Months to <18 years of age with moderate-to-severe atopic dermatitis.

This study will last about 68 weeks and may include up to 16 planned visits. If participating in the optional extension as well, the study will last approximately 1 additional year for a total of up to 116 weeks and may include up to 29 scheduled visits.

ELIGIBILITY:
Inclusion Criteria:

* Received treatment in Study KGBI and have adequately completed the study treatments and last visit of study KGBI, including any applicable systemic AD treatment washout.
* For female participants of childbearing potential, highly effective contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Developed an serious adverse events (SAE) during their participation in parent study KGBI deemed related to lebrikizumab, which in the opinion of the investigator or of the medical monitor could indicate that continued treatment with lebrikizumab may present an unreasonable risk for the participant.
* Developed an AE during their participation in the study KGBI that was deemed related to lebrikizumab and led to study treatment discontinuation, which in the opinion of the investigator or of the medical monitor could indicate that continued treatment with lebrikizumab may present an unreasonable risk for the participant.
* Met the criteria for permanent study intervention discontinuation in study KGBI, if deemed related to lebrikizumab or led to investigator- or sponsor-initiated withdrawal of participant from the study (for example, noncompliance, inability to complete study assessments, etc.)

Note: If study KGBI is still blinded at the time of rollover to study KGBJ, conditions deemed related to the study treatment will be considered related to lebrikizumab.

* Are pregnant or breastfeeding or are planning to become pregnant or breastfeed during the study.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 310 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Discontinued From Study Treatment due to Adverse Events (AEs) | Baseline through Week 52

SECONDARY OUTCOMES:
Percentage of Participants with an Investigator's Global Assessment (IGA) Score 0 or 1 and a Reduction ≥2 Points from Baseline of Study KGBI by Visit in Study KGBJ | Baseline to Week 52
Percentage of Participants Achieving Eczema Area and Severity Index (EASI-75) (≥75% Reduction in EASI Score) from Baseline of Study KGBI by Visit in Study KGBJ | Baseline to Week 52
Percentage of Participants Achieving EASI-90 (≥90% Reduction in EASI Score) from Baseline of Study KGBI by Visit in Study KGBJ | Baseline to Week 52
Percentage of Participants with a Pruritus Numeric Rating Scale (NRS) of ≥4 points at Baseline of Study KGBI who Achieve a ≥4-point Reduction from Baseline of Study KGBI by Visit in Study KGBJ | Baseline to Week 52
Percentage Change from Baseline of Study KGBI by Visit in Study KGBJ in Pruritus NRS Score | Baseline, Week 52
Percentage Change from Baseline of Study KGBI by Visit in Study KGBJ in SCORing Atopic Dermatitis (SCORAD) | Baseline, Week 52
Percentage Change from Baseline of Study KGBI by Visit in Study KGBJ in EASI | Baseline, Week 52
Change from Baseline of Study KGBI by Visit in Study KGBJ in EASI | Baseline, Week 52
Change from Baseline of Study KGBI by Visit in Study KGBJ in Body Surface Area (BSA) | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (94):
- United States (21):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Research Trials, North Little Rock, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - Integrative Skin Science and Research - Location 2, Sacramento, California
  - UConn Health, Farmington, Connecticut
  - Solutions Through Advanced Research, Jacksonville, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Allergy and Asthma Specialist, Owensboro, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Respiratory Medicine Research Institute of Michigan, PLC, Ypsilanti, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Wright State Physicians, Fairborn, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (7):
  - Instituto de Neumonología Y Dermatología, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Psoriahue, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Fundacion Cidea, Buenos Aires, Buenos Aires F.D.
  - Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - Fundación Respirar, Buenos Aires
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Cornerstone Dermatology, Coorparoo, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
- Brazil (8):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Pesquisare Saude, Santo André, São Paulo
  - Clinica de Alergia Martti Antila, Sorocaba, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
- Canada (2):
  - Dermatology Research Institute, Calgary, Alberta
  - DermEdge Research, Mississauga, Ontario
- Czechia (2):
  - Detska nemocnice FN Brno, Brno, Brno-město
  - Fakultni nemocnice Bulovka, Prague, Praha 8
- France (4):
  - Hôpitaux Drôme Nord - Romans, Romans-sur-Isère, Drôme
  - Hôpital Saint Vincent-de-Paul, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes, Loire-Atlantique
  - CHU de Toulouse - Hopital Larrey, Toulouse, Midi-Pyrénées
- Germany (5):
  - Rosenpark Research GmbH, Darmstadt, Hesse
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim, Bad Bentheim, Niedersach
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
- Japan (12):
  - Fujita Health University, Toyoake, Aichi-ken
  - Fukuyama City Hospital, Fukuyama, Hiroshima
  - Asahikawa Medical College Hospital, Asahikawa, Hokkaido
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - Ina Central Hospital, Ina, Nagano
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Dermatology and Ophthalmology Kume Clinic, Sakai, Osaka
  - Enomoto Clinic, Kumagaya, Saitama
  - Sugamo Sengoku Dermatology, Toshima City, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Okayama City General Medical Center Okayama City Hospital, Okayama
- Mexico (9):
  - Instituto Dermatologico de Jalisco, Zapopan, Jalisco
  - Hospital de Jesús Nazareno, Mexico City, Mexico City
  - Trials in Medicine, Mexico City, Mexico City
  - Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico City
  - PanAmerican Clinical Research - Cuernavaca, Cuernavaca, Morelos
  - Eukarya PharmaSite, Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Arké SMO S.A de C.V, Veracruz
- Poland (4):
  - Centrum Medyczne Evimed, Warsaw, Masovian Voivodeship
  - Diamond Clinic, Krakow, Małopolski
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - DERMED Centrum Medyczne Sp. z o.o., Lodz, Łódź Voivodeship
- Spain (10):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona [Barcelona]
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las, Las Palmas
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - CHOP-Centro De Especialidades De Mollabao, Pontevedra, Pontevedra [Pontevedra]
  - Hospital de Manises, Manises, València
  - Grupo Pedro Jaén, Madrid
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Taiwan (6):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Chung Shan Medical University Hospital, Taichung, Taichung
  - National Taiwan University Hospital - Hsinchu branch, Hsinchu
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study to Assess the Long-Term Safety and Efficacy of Lebrikizumab (LY3650150) in Participants 6 Months to <18 Years of Age With Moderate-to-Severe Atopic Dermatitis (ADorable-2) — https://trials.lilly.com/en-US/trial/389036